CLINICAL TRIAL: NCT02001389
Title: A Phase 1, Open-Label, Multiple Ascending Dose, [18F]MNI-659 PET-Imaging Study to Evaluate PDE10A Occupancy After Dosing With EVP-6308 in Healthy Subjects
Brief Title: Study of EVP-6308 to Assess the Dose- and Concentration-dependent Displacement of [18F]MNI-659 by EVP-6308
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EVP-6308-002
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Last update posted 2014-10-10 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Enzyme occupancy; Positron emission tomography (PET); Phosphodiesterase 10 inhibitor

ARMS (4):
- EVP-6308; Arm 1 (Experimental): low dose, Capsule, Twice Daily, Day 1 through Day 3
  Interventions: Drug: EVP-6308
- EVP-6308; Arm 2 (Experimental): low intermediate dose, Capsule, Twice Daily, Day 1 through Day 3
  Interventions: Drug: EVP-6308
- EVP-6308; Arm 3 (Experimental): high intermediate dose, Capsule, Once Daily, Day 1 through Day 3
  Interventions: Drug: EVP-6308
- EVP-6308; Arm 4 (Experimental): high dose, Capsule, Once Daily, Day 1 through Day 3
  Interventions: Drug: EVP-6308

INTERVENTIONS:
Drug: EVP-6308 — Arms 1, 2, 3, 4

SUMMARY:
This is an open-label, single-arm, multiple ascending dose Phase I study to assess the dose- and concentration-dependent displacement of [18F]MNI-659 [a PET tracer targeting phosphodiesterase 10 (PDE10)] by EVP-6308.

ELIGIBILITY:
Inclusion Criteria:

• Healthy male or female volunteers, 18 to 50 years of age

Exclusion Criteria:

* Clinically significant abnormalities on physical examination, medical history, ECG , vital signs, laboratory values, or unstable medical or psychiatric illness
* Any disorder that may interfere with drug absorption.
* Clinically significant allergy or sensitivity to medications Positive test for human immunodeficiency virus (HIV) antibodies, Hepatitis B surface antigen, or Hepatitis C antibody.
* Pregnant or breast feeding.
* History of exposure to any radiation >15 mSv/year (e.g., occupational or radiation therapy) over the past year.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2013-10; Primary Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Target occupancy of [18F]MNI-659. | Baseline and Day 3
  Change in binding potential.

SECONDARY OUTCOMES:
Safety of EVP-6308 as assessed by adverse events, vital signs, clinical laboratory tests, C-SSRS, and electrocardiogram (ECG). | Baseline to Day 4 or Early Termination
  The following will be evaluated: clinical laboratory evaluations (chemistry, hematology, coagulation and urinalysis), physical examination, directed neurological examination, vital signs, orthostatic blood pressure, 12-lead ECG, and assessment for suicidality. Adverse events and concomitant medications will be collected from the time of signing the informed consent.
Pharmacokinetics of EVP-6308 and EVP-6308 N-oxide. | Day 3
  Pharmacokinetic parameters to be determined include Cmax, Tmax, t1/2, and CL/F.

CONTACTS AND LOCATIONS:
Locations (1):
- New Haven, Connecticut, United States